CLINICAL TRIAL: NCT06925789
Title: Influence of Standardized Peri-operative Anesthetic and Analgesic Care on the Outcome of Patients Undergoing Hip Fracture Surgeries
Brief Title: Influence of Standardized Perioperative Anesthetic, Analgesic Care on Outcome of Patients Undergoing Hip Fracture Surgeries
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: We changed the study design.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Shubha Srinivasareddy, Assistant Professor of Anesthesia and Peri-operative care, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 25751
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-06

CONDITIONS: Fractures, Hip; Local Anesthesia; Geriatric; Nerve Block
Keywords: Hip Fracture; Nerve blocks; Geriatric; Local anesthesia; Post operative outcomes
MeSH Terms: conditions — Hip Fractures | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Local anesthesia to treat hip fracture in geriatric patients (Experimental)
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — The nerve block is performed when the patients are admitted to the hospital with diagnosed hip fractures. And another nerve block with catheter is performed for post-operative pain control in geriatric population with 0.25% Ropivacaine 30mls.

SUMMARY:
The purpose of this voluntary research study is to clarify whether or not a single injection nerve block done before surgery and after surgery nerve block catheter can effectively enhance recovery in elderly hip fracture patients in terms of reduced delirium, reduced length of stay and improved surgical and anesthesia outcomes. Delirium is a serious change in mental abilities. It results in confused thinking and a lack of awareness of someone's surroundings. The disorder usually comes on fast - within hours or a few days. Prolonged hospital stay is one of the risk factors for onset of delirium.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing anesthesia for hip fracture surgery.
2. Patients with fracture neck of femur fractures.
3. Geriatric patients. (65 years and older)

Exclusion Criteria:

1. Non-fracture hip patients
2. non-geriatric patients. (Below 65 years old)
3. Patients not able to consent themselves
4. Non- English-speaking patients

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain Control | up to 48 hours post hospital admission.
  Pain control is determined by the Likert pain scale, where 0 is no pain and 10 as severe pain
Opioid Use | up to 48 hours post hospital admission.
  Identification of opioid use via the EMR, Opioids usage is measured at as number of morphine equivalents during the hospital admission.

SECONDARY OUTCOMES:
Delirium score | up to 48 hours post hospital admission.
  Delirium score is calculated using the FLACC score, where FLACC score of 0 is relaxed and comfortable and FLACC score of 7-10 is severe delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Shubha Srinivasareddy, MD, Principal Investigator — Penn State Health

IPD SHARING:
Plan to Share IPD: No